CLINICAL TRIAL: NCT04284917
Title: Evaluate the Long Term Effectiveness & Safety of the Use of Carglumic Acid (Carbaglu®) in Patients With Propionic Acidemia (PA) or Methylmalonic Acidemia (MMA).
Brief Title: Long-term Efficacy of Carglumic Acid in Organic Acidemia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201810033MIPB
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Propionic Acidemia (PA) , Methylmalonic Acidemia (MMA)
Keywords: Carglumic Acid (Carbaglu®)
MeSH Terms: conditions — Propionic Acidemia; Methylmalonic acidemia | interventions — carglumic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receive Carglumic Acid (Experimental): Experimental Case_ Carglumic Acid
  Interventions: Drug: Carglumic Acid (Carbaglu®)

INTERVENTIONS:
Drug: Carglumic Acid (Carbaglu®) — A. Study period: 36 months; treatment period: 12 months.
  B. Patients will receive Carglumic Acid (Carbaglu®) 50 mg/kg/day in addition to standard therapy (protein restricted diet, L-carnitine, metronidazole and vitamin B12).
  C. Patients need to regularly come back for follow up examination on Day 0, month 3, month 6, and month 12.
  D. Patients should report any adverse event that occur during treatment period.
  E. Patients' number of emergency visits due to hyperammonemia, ammonia level, acylcarnitine, urinary organic acid analysis, plasma amino acid analysis and methylmalonic acid will be recorded during treatment period.

SUMMARY:
Evaluate the Long Term Effectiveness & Safety of the use of Carglumic Acid (Carbaglu®) in Patients with Propionic Acidemia (PA) or Methylmalonic Acidemia (MMA).

DETAILED DESCRIPTION:
Study procedures:

A. Study period: 36 months; treatment period: 12 months.

B. Patients will receive Carglumic Acid (Carbaglu®) 50 mg/kg/day in addition to standard therapy (protein restricted diet, L-carnitine, metronidazole and vitamin B12).

C. Patients need to regularly come back for follow up examination on Day 0, month 3, month 6, and month 12.

D. Patients should report any adverse event that occur during treatment period.

E. Patients' number of emergency visits due to hyperammonemia, ammonia level, acylcarnitine, urinary organic acid analysis, plasma amino acid analysis and methylmalonic acid will be recorded during treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. PA or MMA confirmed using the following criteria:

   * PA confirmed by the measurement of acylcarnitine profile, urine organic acid, measurement of propionyl Co-A carboxylase in leukocytes or cultured fibroblasts or by DNA molecular testing of PCCA (Propionyl CoA Carboxylase, Alpha Polypeptide) or PCCB (propionyl CoA carboxylase, beta polypeptide) gene
   * MMA confirmed by the measurement of acylcarnitine profile, urine organic acid, measurement of methymalonyl Co-A mutase in culture fibroblasts or DNA molecular testing of mutgene.
2. Male or female Children of 18 years old or less.
3. Had experienced Hyperammonemia(NH3 ≧100 uM) before.
4. Not participating in any other clinical trial in the previous 30 days

Exclusion Criteria:

1. Patients with other organic acidemia or any other cause of hyperammonemia
2. Patient receiving other investigational therapy for PA or MMA
3. Patient with PA or MMA and other inherited genetic conditions or congenital anomalies
4. Past history of hypersensitivity or drug allergy to Carbaglu®

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Number of emergency visits due to hyperammonemia within 12 months period | 12 months
  Adverse Events

SECONDARY OUTCOMES:
Time to first visit to the ER due to hyperammonemia from starting the treatment | 12 months
  Adverse Events
Assessment of Plasma ammonia level | Baseline,3,6,9 and 12,months after receiving Carbaglu.
  Plasma ammonia level over the study treatment period.
Number of days of hospitalization | 12 months
  Number of days of hospitalization during study treatment period.
Assessment of Acylcarnitine level | Baseline,3,6,9 and 12,months after receiving Carbaglu.
  Acylcarnitine level for all patients
Assessment of urine organic acid level | Baseline,3,6,9 and 12,months after receiving Carbaglu.
  Measuring urine organic acid level for both diseases.
Assessment of Plasma aminoacids' level | Baseline,3,6,9 and 12,months after receiving Carbaglu.
  Measuring Plasma aminoacids' level for both diseases.
Assessment of Methylmalonic acid level | Baseline,3,6,9 and 12,months after receiving Carbaglu.
  Measuring Methylmalonic acid level for both diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Ni-Chung Lee, M.D., Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan